CLINICAL TRIAL: NCT03392025
Title: Effects of Flaxseed Consumption, Alone and in Combination With the Mediterranean-like Diet, on Vascular Endothelial Function and Some Biochemical Indicators Related to Atherosclerosis in Patients With Coronary Artery Disease
Brief Title: Flaxseed Consumption, Alone and in Combination With the Mediterranean-like Diet, on Some Indicators Related to Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javad Nasrollahzadeh (Other)
Responsible Party: Sponsor-Investigator, Javad Nasrollahzadeh, Director, Shahid Beheshti University
Organization: Shahid Beheshti University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 651
Record Dates: First submitted 2017-12-07; First posted 2018-01-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Linseed Oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flaxseed (Active Comparator): Daily consumption of 30 grams flaxseed for 3 months
  Interventions: Other: Flaxseed
- Flaxseed and the Mediterranean-like diet (Active Comparator): Daily consumption of 30 grams flaxseed in adjunct to the Mediterranean-like diet for 3 months
  Interventions: Other: Flaxseed; Other: the Mediterranean-like diet
- Placebo (Placebo Comparator): Daily consumption of Placebo for 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: Flaxseed — Daily consumption of 30 grams flaxseed in adjunct to medical treatment for 3 months
  Arms: Flaxseed; Flaxseed and the Mediterranean-like diet
Other: the Mediterranean-like diet — Weekly Mediterranean-like diet menu in adjunct to medical treatment for 3 months
  Arms: Flaxseed and the Mediterranean-like diet
Dietary Supplement: Placebo — Daily consumption of one capsule of wheat fiber as placebo in adjunct to medical treatment for 3 months
  Arms: Placebo

SUMMARY:
Flaxseed consumption has beneficial effects on cardiovascular risk factors. In addition, the benefit of the Mediterranean-like diet in primary and secondary prevention of cardiovascular diseases has been shown.The purpose of this study is to investigate the effects of flaxseed consumption, alone and in combination with the Mediterranean-like diet, in adjunct to conventional medical treatment, in improving vascular endothelial function, plasma lipid profile and high sensitivity c-reactive protein of coronary artery disease (CAD) patients.

DETAILED DESCRIPTION:
A randomized placebo controlled clinical trial will be conducted in Rajaie Cardiovascular Center in Tehran, Iran. After review of the inclusion and exclusion criteria and explanation of the design of the study, written consent form will be completed. The participants are 81 eligible coronary artery disease patients, aged 20-75 years. Intervention groups will be received 30 g/d flaxseed, alone, or with weekly Mediterranean-like diet menu and control group will be received capsules of wheat fiber as placebo for 3 months. Vascular endothelial function will be evaluated through measurement of flow mediated dilatation (FMD) in brachial artery and carotid intima-media thickness (c-IMT) via ultrasound sonography and plasma level of asymmetric di-methyl arginine (ADMA). Fasting blood sample will be taken to measure malondialdehyde (MDA), lipid profile, high sensitive C-reactive protein and inflammatory cytokines (Interleukine-6 [IL-6] and Tumor Necrosis Factor-a [TNF-a]).

ELIGIBILITY:
Inclusion Criteria:

1. coronary artery disease patients (more than 50% blockage in coronary arteries) needed angioplasty with stent
2. willing to participation in the study

Exclusion Criteria:

1. cigarette Smoking
2. continuous consumption of any antioxidant supplement such as vitamin E, vitamin C and Selenium in last month
3. consumption of flaxseed or any omega-3 supplement at the beginning of the study
4. َadvanced renal disease
5. unwillingness to continuance
6. any change in disease treatment plan such as change in type and dose of lipid lowering drugs or surgical operation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation (FMD) | 3 month
  Change in dilatation of the brachial artery from baseline at 3 month

SECONDARY OUTCOMES:
plasma level of high sensitive C reactive protein (hs-CRP) | 3 month
  change in plasma level of high sensitive C reactive protein (hs-CRP) from baseline at 3 month
plasma lipid profile | 3 month
  change in plasma level of lipid profile from baseline at 3 month
carotid intima-media thickness (c-IMT) | 3 month
  change in carotid intima-media thickness from baseline at 3 month
asymmetric di-methyl arginine (ADMA) | 3 month
  change in plasma level of assymetric di-methyl arginine from baseline at 3 month

OTHER OUTCOMES:
plasma levels of Interleukine-6 (IL-6) | 3 month
  change in plasma levels of IL-6 from baseline at 3 month
plasma levels of malondialdehyde (MDA) | 3 month
  change in plasma levels of MDA from baseline at 3 month
plasma levels of Tumor Necrosis Factor-alfa (TNF-a) | 3 month
  change in plasma levels of TNF-a from baseline at 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nasrollahzadeh, Ph.D, Study Chair — Department of Clinical Nutrition and Diet Therapy, National Nutrition and Food Technology Research Institute, Faculty of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences; Javad Nasrollahzadeh, Ph.D, Study Director — Department of Clinical Nutrition and Diet Therapy, National Nutrition and Food Technology Research Institute, Faculty of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences; Nafiseh Khandouzi, Ph.D student, Principal Investigator — Department of Clinical Nutrition and Diet Therapy, National Nutrition and Food Technology Research Institute, Faculty of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences
Locations (1):
- Rajaie Cardiovascular, Medical & Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cassani RS, Fassini PG, Silvah JH, Lima CM, Marchini JS. Retraction Note: Impact of weight loss diet associated with flaxseed on inflammatory markers in men with cardiovascular risk factors: a clinical study. Nutr J. 2016 Jun 7;15(1):59. doi: 10.1186/s12937-016-0165-x. No abstract available. PMID 27267967
- [Background] Widmer RJ, Flammer AJ, Lerman LO, Lerman A. The Mediterranean diet, its components, and cardiovascular disease. Am J Med. 2015 Mar;128(3):229-38. doi: 10.1016/j.amjmed.2014.10.014. Epub 2014 Oct 15. PMID 25447615
- [Background] Ros E, Martinez-Gonzalez MA, Estruch R, Salas-Salvado J, Fito M, Martinez JA, Corella D. Mediterranean diet and cardiovascular health: Teachings of the PREDIMED study. Adv Nutr. 2014 May 14;5(3):330S-6S. doi: 10.3945/an.113.005389. Print 2014 May. PMID 24829485
- [Background] Bloedon LT, Balikai S, Chittams J, Cunnane SC, Berlin JA, Rader DJ, Szapary PO. Flaxseed and cardiovascular risk factors: results from a double blind, randomized, controlled clinical trial. J Am Coll Nutr. 2008 Feb;27(1):65-74. doi: 10.1080/07315724.2008.10719676. PMID 18460483
- [Background] Fuentes F, Lopez-Miranda J, Sanchez E, Sanchez F, Paez J, Paz-Rojas E, Marin C, Gomez P, Jimenez-Pereperez J, Ordovas JM, Perez-Jimenez F. Mediterranean and low-fat diets improve endothelial function in hypercholesterolemic men. Ann Intern Med. 2001 Jun 19;134(12):1115-9. doi: 10.7326/0003-4819-134-12-200106190-00011. PMID 11412051
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Murie-Fernandez M, Irimia P, Toledo E, Martinez-Vila E, Buil-Cosiales P, Serrano-Martinez M, Ruiz-Gutierrez V, Ros E, Estruch R, Martinez-Gonzalez MA; PREDIMED Investigators. Carotid intima-media thickness changes with Mediterranean diet: a randomized trial (PREDIMED-Navarra). Atherosclerosis. 2011 Nov;219(1):158-62. doi: 10.1016/j.atherosclerosis.2011.06.050. Epub 2011 Jul 6. PMID 21802081
- [Background] Marin C, Ramirez R, Delgado-Lista J, Yubero-Serrano EM, Perez-Martinez P, Carracedo J, Garcia-Rios A, Rodriguez F, Gutierrez-Mariscal FM, Gomez P, Perez-Jimenez F, Lopez-Miranda J. Mediterranean diet reduces endothelial damage and improves the regenerative capacity of endothelium. Am J Clin Nutr. 2011 Feb;93(2):267-74. doi: 10.3945/ajcn.110.006866. Epub 2010 Dec 1. PMID 21123460